CLINICAL TRIAL: NCT01914887
Title: A Phase I/IIa Clinical Trial to Evaluate Safety and Efficacy of Adipose Tissue-derived Mesenchymal Stem Cells (ASC) on Induction to Remission in Ulcerative Colitis
Brief Title: Allogeneic Adipose Tissue-derived Mesenchymal Stem Cells for the Induction of Remission in Ulcerative Colitis
Acronym: ALOASCU
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: Fundacion para la Investigacion Biomedica del Hospital Universitario la Paz (Other); Ministry of Health, Spain (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLPDIG-2010-01; 2010-023798-20 (EudraCT Number)
Record Dates: First submitted 2013-07-18; First posted 2013-08-02 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-07

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; Inflammatory Bowel Disease; Mesenchymal stem cells
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- allogeneic ASCs (Experimental): Treatment consists in a cell suspension (5 million cells/mL) in aseptic buffered solution containing human expanded adipose-derived stem cells (eASCs) of allogeneic origin in disposable vials with no preservative agents. The cells will be given in different sites within the affected colonic submucosa at a total dose of 60 million cells with the use of a colonoscope.
  Interventions: Drug: Allogeneic adipose tissue-derived mesenchymal stem cells

INTERVENTIONS:
Drug: Allogeneic adipose tissue-derived mesenchymal stem cells — The cells will be given in different sites within the affected colonic submucosa at a total dose of 60 million cells with the use of a colonoscope.
  Other Names: Cx-601 (company code)

SUMMARY:
The aims of our study are to evaluate the feasibility and safety of endoscopic injection of adipose tissue-derived mesenchymal stem cells in human subjects with moderate active ulcerative colitis, assessing the absence of adverse events associated to the investigational drug, and to evaluate the efficacy of the treatment to induce remission of moderate active ulcerative colitis, by improvements in disease activity index, quality of life index, and endoscopic index.

DETAILED DESCRIPTION:
Mesenchymal stem cells (MSC) may be a therapeutic option in diseases associated with severe inflammation or auto-immune diseases, due to their immunomodulatory and anti-inflammatory properties. A number of clinical trials are being conducted worldwide testing th efficacy of MSC, mainly isolated from bone marrow, for different conditions, such as Graft Versus host Disease, refractory Crohn's Disease, ischemic stroke, acute myocardial infarction, type I Diabetes Mellitus, or Chronic Obstructive Pulmonary Disease. Usually, the route of administration of the cells in these studies is intravenous. Local injection of MSC for fistulizing Crohn's Disease has proven efficacious. Endoscopy is a routinary technique for the evaluation of gastrointestinal and colonic conditions. The purpose of our study is to evaluate safety and efficacy of the intracolonic injection by using a colonoscope of allogeneic adipose tissue-derived MSC in patients with moderate active ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex aged 18 years and older
* Signed informed consent
* Patients with ulcerative colitis diagnosed at least 6 months earlier in accordance with usual criteria
* Left-sided colitis with moderate activity defined by a modified Truelove-Witts score between 11 and 21, and with no response to 4 weeks of treatment with oral and/or topical 5-aminosalicylates
* Negative pregnancy test for women of childbearing potential (from menarche to menopause) using consistently and correctly highly effective (i.e. less than 1% failure rate per year) methods of birth control

Exclusion Criteria:

* Mental disability that impedes adequate understanding of the study and of the associated procedures
* Extensive colitis
* Patients with an impaired general state which requires, according to the investigator judgment, immediate treatment with corticosteroids and/or anti-Tumor Necrosis Factor (TNF) and/or surgery
* Patients that fulfill criteria of corticodependency and in ongoing treatment with corticosteroids
* Patients with previous colectomies
* Known history of alcohol or other addictive substances abuse
* History of malignant disease - Patients having participated in clinical trials with any investigational drug within 6 months prior to enrolment in this study
* Patients with known allergies to penicillin, gentamicin, aminoglycosides, human serum albumin (HSA), Dulbecco's modified Eagle medium (DMEM), or materials of bovine origin
* Pregnant or breastfeeding women
* Presence of severe concomitant diseases
* Patients with suspicion of Crohn?s enterocolitis, indeterminate colitis, ischaemic colitis, radiation colitis, diverticular disease associated colitis, or microscopic colitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2013-06; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Safety | Up to 12 weeks
  Evaluation of the presence of any event that could be considered adverse event, especially if it can be attributed to the investigational drug. Physical exam, vital signs, and laboratory tests (hemogram, biochemistry, coagulation, and cytokines) will be performed at 0, 9-10 days, and 4, 8, and 12 weeks.

SECONDARY OUTCOMES:
Efficacy: Change from Baseline in Modified Truelove-Witts score | Up to 12 weeks
  Remission will be considered if it descends below 11, and response if it diminishes at least 30%. Modified Truelove-Witts score will be evaluated at 0, 4, 8, and 12 weeks.
Efficacy: Change from Baseline in Quality of Life index, Inflammatory Bowel Disease Questionnaire (IBDQ-32) | Up to 12 weeks
  Response will be considered if it improves at least 30%. IBDQ-32 will be evaluated at 0, 4, 8, and 12 weeks.
Efficacy: Change from baseline in Mayo endoscopic index. | 8 weeks
  Remission will be considered if reaches 0 points and response if the score diminishes. Endoscopy will be performed at 0 and 8 weeks.
Change from Baseline in C Reactive Protein | Up to 12 weeks
  C Reactive Protein will be evaluated at 0, 9-10 days, and 4, 8, 12 weeks.
Change from Baseline in fecal calprotectin | Up to 12 weeks
  Fecal calprotectin will be evaluated at 0, 4, 8, and 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Dolores Martin Arranz, MD, Principal Investigator — Gastroenterology Department
Locations (1):
- Hospital Universitario La Paz, Madrid, Spain

REFERENCES:
- [Background] Garcia-Gomez I, Elvira G, Zapata AG, Lamana ML, Ramirez M, Castro JG, Arranz MG, Vicente A, Bueren J, Garcia-Olmo D. Mesenchymal stem cells: biological properties and clinical applications. Expert Opin Biol Ther. 2010 Oct;10(10):1453-68. doi: 10.1517/14712598.2010.519333. PMID 20831449
- [Background] Duijvestein M, Vos AC, Roelofs H, Wildenberg ME, Wendrich BB, Verspaget HW, Kooy-Winkelaar EM, Koning F, Zwaginga JJ, Fidder HH, Verhaar AP, Fibbe WE, van den Brink GR, Hommes DW. Autologous bone marrow-derived mesenchymal stromal cell treatment for refractory luminal Crohn's disease: results of a phase I study. Gut. 2010 Dec;59(12):1662-9. doi: 10.1136/gut.2010.215152. Epub 2010 Oct 4. PMID 20921206
- [Background] van Deen WK, Oikonomopoulos A, Hommes DW. Stem cell therapy in inflammatory bowel disease: which, when and how? Curr Opin Gastroenterol. 2013 Jul;29(4):384-90. doi: 10.1097/MOG.0b013e328361f763. PMID 23666365